CLINICAL TRIAL: NCT00438009
Title: A Phase I, Open Label, Cohort Study of Two Doses of Cavatak (Coxsackievirus Type A21) Given Intratumourally in Stage IV Melanoma Patients.
Brief Title: A Safety Study of Two Intratumoural Doses of Coxsackievirus Type A21 in Melanoma Patients (PSX-X03)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Viralytics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: V937-003; PAH HREC identifier 2006/49; PSX-X03 (Other: Viralytics Study ID)
Record Dates: First submitted 2007-02-19; First posted 2007-02-21 (Estimated); Last update posted 2019-07-01 (Actual); Status verified 2019-06

CONDITIONS: Stage IV Melanoma
Keywords: coxsackievirus type a21; oncolytic virus; melanoma
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAVATAK (Experimental)
  Interventions: Drug: Coxsackievirus A21

INTERVENTIONS:
Drug: Coxsackievirus A21 — Two doses of drug, separated by 48 hours
  Other Names: CAVATAK

SUMMARY:
The purpose of the study is to determine the safety and tolerability of two doses of Coxsackievirus A21, administered 48 hours apart into a superficial melanoma tumour.

Injected and non-injected tumours will be observed regarding change in tumour size.

Coxsackievirus A21 (CVA21) is a naturally occurring virus, that is known to cause self limiting upper respiratory infections. CVA21 has been shown in cell culture to infect and kill human melanoma cancer cell lines. This property of CVA21 is due to the specific receptors CVA21 uses in order to attach to, and infect a cell. The 2 receptors CVA21 uses to infect a cell are Intracellular Adhesion Molecule 1 (ICAM-1) and Decay Accelerating Factor. Both of these surface proteins are expressed on melanoma cell lines as well as human melanoma tumours. Animal models of human melanoma tumours have demonstrated that CVA21 injection either intratumour or intravenous causes infection in the tumours, resulting in reduction of tumour size and growth.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 18 years of age.
* One subcutaneous melanoma metastatic deposit, 2.0 to 5.0 cm in diameter, accessible to 3mm punch biopsy and injection, may be tumour infiltrated lymph node.
* Melanoma stage IV.
* 3mm punch biopsy of the selected tumour must be expressing ICAM-1 and DAF.
* Absence of circulating antibodies to CVA21 (titre < 1:16)
* Patients must have adequate hematological, renal and hepatic function
* Failed or refused standard treatment (s)
* Patients are able and willing to provide signed/informed consent to participate in the study.
* Fertile males and females must agree to the use of adequate form of contraception, eg. Condoms for males
* Negative pregnancy test is required for female patients of child bearing potential.

Exclusion Criteria:

* Mucosal or ocular tumour
* Presence of CNS tumour
* Radiotherapy to the injection tumour site.
* Prior local radiotherapy without subsequent nodule progression
* Chemotherapy within 4 weeks of screening visit.
* ECOG score greater than 1.
* Life expectancy less than 3 months.
* Pregnancy or breast feeding.
* Primary or secondary immunodeficiency, including immuno-suppressive doses of corticosteroids (prednisolone greater than 7.5 mg/day, or other immuno-suppressive drugs such as cyclosporine, azothioprine, interferons, within the 4 weeks prior to screening visit.
* Positive serology for HIV, Hepatitis B virus or Hepatitis C virus
* Full dose anticoagulation, or a history of bleeding diathesis, or history of difficult to control bleeding in the month before screening visit.
* Previous splenectomy.
* Presence of uncontrolled infection.
* Presence of unstable neurological disease
* Any uncontrolled medical condition that in the opinion of the Investigator is likely to place the patient at unacceptable risk during the study or reduce their ability to complete the study
* Participation in another study requiring administration of an investigational drug or biological agent within the last 4 weeks prior to screening visit.
* Known allergy to treatment medication or excipients
* Any other medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-05-16 (Actual); Primary Completion 2009-08-28 (Actual); Study Completion 2009-08-28 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of two doses of Coxsackievirus A21 administered intratumourally. | Days 1, 3, 6, 8, 10, 13, 17, 24, 38, 52, 87

SECONDARY OUTCOMES:
To determine clinical response of the injected tumour | Days 24, 52, 87
To determine clinical response in non-injected tumours using RECIST criteria | 3 months
Time course and quantify CVA21 viremias | 3 months
Determine time course to elimination of CVA21 | 3 months
Determine time course, frequency as well as quantify the development of anti-CVA21 antibodies | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Alexandra Hospital, Brisbane, Queensland, Australia

REFERENCES:
- [Background] Shafren DR, Au GG, Nguyen T, Newcombe NG, Haley ES, Beagley L, Johansson ES, Hersey P, Barry RD. Systemic therapy of malignant human melanoma tumors by a common cold-producing enterovirus, coxsackievirus a21. Clin Cancer Res. 2004 Jan 1;10(1 Pt 1):53-60. doi: 10.1158/1078-0432.ccr-0690-3. PMID 14734451
- [Background] Au GG, Lindberg AM, Barry RD, Shafren DR. Oncolysis of vascular malignant human melanoma tumors by Coxsackievirus A21. Int J Oncol. 2005 Jun;26(6):1471-6. doi: 10.3892/ijo.26.6.1471. PMID 15870858
- See also: Sponsor Website — http://viralytics.com